CLINICAL TRIAL: NCT04983602
Title: The Effectiveness of a Physiotherapy Led Community Based Intervention at Reducing Adverse Outcomes in Older Adults Discharged From the Emergency Department: A Pilot Feasibility Randomized Controlled Trial
Brief Title: Physiotherapy Led Community Intervention for Older Adults Discharged From the Emergency Department
Acronym: EDPLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: University Hospital of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDPLUS
Record Dates: First submitted 2021-06-23; First posted 2021-07-30 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Old Age; Debility; Health Services for the Aged
Keywords: older adults; geriatric medicine; integrated care; emergency department; feasibility
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be unaware if the participant was in usual care, comprehensive geriatric assessment arm or the ED PLUS arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care Control group (No Intervention): The usual care control group receives conventional care in the Emergency Department (ED) or Acute Medical Assessment Unit (AMAU)The comparison group will receive routine care as would be usual in the ED or AMAU. Currently there is no dedicated team to perform CGA in the ED and AMAU at UHL with ad hoc allied health assessment available only at the discretion of the referring ED doctor or medical team. This process will be continued during the study and will be documented. The participants in this group will under baseline data collection prior to randomisation and follow up.
- Comprehensive Geriatric assessment arm (Experimental): The intervention will comprise initially of a detailed interdisciplinary assessment and intervention by one or more members of the dedicated geriatric team. The team (consisting of a geriatric specialist registrar, specialist geriatric nurse, senior pharmacist, senior physiotherapist, senior occupational therapist, and senior medical social worker) in both ED and AMAU will assess all participants in the intervention group and perform CGA. Potential participants will be approached regarding trial recruitment post ED triage thereby ensuring rapid assessment shortly after hospital arrival by the teams in both AMAU and in ED.
  Interventions: Other: Comprehensive Geriatric Assessment arm
- EDPLUS arm (Experimental): The ED PLUS intervention will comprise initially of a detailed interdisciplinary assessment and intervention by one or more members of the dedicated geriatric team. The team in both ED and AMAU will assess all participants in the intervention group and perform CGA. Potential participants will be approached regarding trial recruitment post ED triage thereby ensuring rapid assessment shortly after hospital arrival by the teams in both AMAU and in ED. Additionally the participants in this arm will undergo a 6 week physiotherapy led intervention in the community involving 3 home visits and weekly telephone support. The intervention will involved assessment of the patients function in terms of strength, balance and mobility. Following assessment the intervention will be aimed at addressing deficits in the function of the participants, review of their medical management by a geriatrician trainee and focusing on self management of their own program.
  Interventions: Other: EDPLUS

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment arm — The intervention will involve a comprehensive geriatric assessment which will be provided by a geriatric doctor, physiotherapist, occupational therapist, social worker, pharmacist and specialist nurse.,
  Arms: Comprehensive Geriatric assessment arm
Other: EDPLUS — EDPLUS involves a 6 week physiotherapy led community based intervention involving 3 home visits and weekly telephone support.
  Arms: EDPLUS arm

SUMMARY:
ED PLUS Emergency Department Discharge Physiotherapy Led Community Service is a pilot feasibility randomized controlled trial investigating the role of an integrated care intervention consisting of comprehensive geriatrics assessment in older adults in the emergency department and a physiotherapy-led community based intervention.

DETAILED DESCRIPTION:
All patients who are aged 65 years and over will be screened using the Identification of Seniors at Risk (ISAR) Tool in the emergency department of a University Teaching Hospital. Those with a score of 2 or above in the ISAR and suitable for discharge home will be randomised. The first treatment arm will undergo geriatric medicine item directed Comprehensive Geriatric Assessment (CGA) from admission to emergency department (ED). The non-treatment arm will under usual patient care. The second treatment arm will undergo geriatric medicine team directed CGA from admission to ED and a physiotherapy led community based 6 week intervention in the patient's home. A dedicated multidisciplinary team of geriatric medicine trainee, occupational therapist, physiotherapist and medical social worker will carry out the assessment. For those randomised to the second treatment arm, a physiotherapist will assess and carry out a 6 week interventions that arise from that assessment and liaise with the patients General Practitioner (GP), medical social worker and other health care professionals. The overall aims of ED PLUS are assess the feasibility of the 6 week physiotherapy led intervention. Feasibility will be determined by the following outcomes:

i) Recruitment rate

ii) Adherence rate

iii) Acceptability of the programme

iv) Retention

v) Incidents

The secondary aims are to improve function, reduce anxiety and depression, improve quality of life and prevent unnecessary ED admission.

ELIGIBILITY:
The inclusion criteria for participants include:

* Adults aged ≥65 years with undifferentiated medical complaints presenting to an ED.
* Medically stable as deemed by the treating physician
* Display a score of ≥2 on the Identification of Seniors at Risk (ISAR) screening tool.
* Be community dwelling
* Be discharged from the ED within 72 hours of index visit.

Exclusion criteria include:

* Individuals under the age of 65 years.
* Have a score of less than 2 on the ISAR.
* Older adults who present with acute myocardial infarction, stroke or non-medical problems e.g. surgical or psychiatric issues.
* Older adults who are medically unstable will be excluded.
* If neither the patient nor carer can communicate in English sufficiently to complete consent or baseline assessment, they will be excluded.
* Older adults who are admitted to hospital from the ED will be excluded.
* Older adults who have a confirmed COVID 19 diagnosis or those with symptoms highly suggestive of COVID 19 will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Functional Decline | 6 weeks post ED visit
  Barthel Index is global measure of functional status with a score from 0-20. A score of 0 is completely dependent, 20 is fully independent.
Functional Decline | 6 months post ED visit
  Barthel Index is global measure of functional status with a score from 0-20. A score of 0 is completely dependent, 20 is fully independent.

SECONDARY OUTCOMES:
Patient Quality of Life | Baseline, 6 weeks post ED visit and 6 months post ED visit
  Patient rated quality of life is determined by the Euro Quality of Life EQ5D. This scale is scored from 0 to 100 where 0 is the worst imaginable health state with 100 being the best imaginable.
Patient satisfaction | Baseline, 6 weeks post ED visit and 6 months post ED visit
  Patient satisfaction is determined by the Patient Satisfaction Survey III Short Form (PSQ18). This is scored from 18 to 90, with 18 being the lowest level of satisfaction to 90 being the best score
Rate of ED representation | Baseline, 6 weeks post ED visit and 6 months post ED visit
  A record of the patient coming back to the ED within 6 weeks and/or 6 months post ED index visit
Rate of Hospital readmission | Baseline,6 weeks post ED visit and 6 months post ED visit
  A record of the patient requiring admission to the hospital within 6 weeks and/or 6 months
Mortality | 6 weeks post ED index visit or 6 months post ED index visit
  A record of the patient having died within 6 weeks or 6 months
Patient Experience Times | 6 weeks
  Exact time of admission or discharge form the ED will be collected at 6 weeks post ED index visit
Number of visits to the family doctor or public health nurse | 6 weeks and 6 months post index ED visit
  Determined by self reported visits to family doctor or public health nurse. This will be a telephone consultation at 6 week and 6 months post ED index visit where patients will be asked if they have visited a family doctor or public health nurse in the previous 6 weeks at the 6 week telephone call, or 6 months at the 6 month telephone call

CONTACTS AND LOCATIONS:
Overall Officials: Rose Galvin, PhD, Principal Investigator — University of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be stored on a data repository after the study analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study protocol will be prepared for publication in an open access journal. The protocol will include the Statistical Analysis plan, detailed descriptions of interventions. It is likely to be published in September 2021
Access Criteria: Supporting information will be available on peer review publications.

REFERENCES:
- [Derived] Conneely M, Leahy S, O'Connor M, Corey G, Gabr A, Saleh A, Okpaje B, O' Shaughnessy I, Synnott A, McCarthy A, Holmes A, Robinson K, Ryan L, Griffin A, Barry L, Trepel D, Ryan D, Galvin R; Ageing Research Centre Public and Patient Involvement (PPI) Panel of older adults. A Physiotherapy-Led Transition to Home Intervention for Older Adults Following Emergency Department Discharge: A Pilot Feasibility Randomised Controlled Trial (ED PLUS). Clin Interv Aging. 2023 Oct 24;18:1769-1788. doi: 10.2147/CIA.S413961. eCollection 2023. PMID 37901478
- See also: Peer reviewed protocol — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-021-00954-5
- See also: shared link — https://rdcu.be/cOGBd